CLINICAL TRIAL: NCT02150629
Title: Investigating Kinematic and Electromyographic Changes After SCI and Their Relation to Clinical and Functional Outcome
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-2011-0257/PB_2016-00228
Record Dates: First submitted 2014-05-13; First posted 2014-05-30 (Estimated); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- SCI patients
- Healthy subjects

SUMMARY:
The study aims at discerning specific gait patterns and elucidating locomotor control of spinal cord injured patients in order to find sensitive kinematic and electromyographic outcome measures that are able to reveal information on underlying mechanisms of normal and aberrant gait control and its recovery over time. These measures may also be used to compare the outcome across different neurological disorders.

ELIGIBILITY:
Inclusion Criteria:

Patients: We will monitor patients who were admitted to the Spinal Cord Injury Center of the University Hospital Balgrist. We will record patients with various aetiologies, grades of impairment and types of spinal cord lesions. Patients need to have minimal voluntary motor capacities: the motor scores of the key muscles according to the ASIA classification (www.asia-spinalinjury.org) should be at least 3 for extensor muscles and 2 for flexor muscles. Written informed consent is required. Control subjects: Healthy subjects, written informed consent.

Exclusion Criteria:

Patients: Comorbidities which influence or inhibit gait or upper-limb motion (e.g. peripheral nerve lesions). Orthostatic problems that greatly impair upright body position. Mental illness, cognitive impairments. Control subjects: neurologic disease, walking disabilities, mental illness, cognitive impairments

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Spinal cord injury patients and healthy control subjects
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change of gait kinematics after spinal cord injury over one year | 1) very acute: 0 - 14 days after injury; 2) acute I: 2 - 4 weeks post-injury; 3) acute II: 4 - 12 weeks post-injury; 4) acute III: 12 - 24 weeks post-injury; 5) chronic: 24 - 48 weeks post-injury

CONTACTS AND LOCATIONS:
Locations (1):
- Balgrist University Hospital, Zurich, Switzerland